CLINICAL TRIAL: NCT06334237
Title: Exploring the Psychosomatic Factors Influencing and Moderating the Efficacy of Holistic Care and Personalized Treatment for Migraine Patients: A Prospective Longitudinal Observational Study
Brief Title: Psychosomatic Factors Influencing the Efficacy of Holistic Care for Migraine
Status: Recruiting | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Y_113_0009
Record Dates: First submitted 2024-02-01; First posted 2024-03-27 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Migraine
Keywords: migraine; holistic care; personalized treatment
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: personalized treatment — According to the condition of each individuals, the study continues their routine clinical care. The study does not offer anything more than a routine clinical care. It is named personalized treatment because the condition of each individual varies, so the doctor may prescribe or offer clinical advice accordingly. .

SUMMARY:
This research project aims at exploring the psychosomatic factors that influence and moderate the efficacy of holistic care and personalized treatment for migraine patients. It is a prospective longitudinal observational study. The project's goal is to understand how physical, psychological, spiritual, and social factors affect the care and treatment outcomes for migraineurs. The study will include participants aged 18 to 65, who meet the International Headache Society's criteria for migraines. It will utilize a range of methodologies including questionnaires, interviews, and medical records to collect data on various factors like lifestyle, psychological state, and social support. The project will assess the effectiveness of treatments, compliance, and other outcomes such as emotional and sleep conditions.

DETAILED DESCRIPTION:
In this study, participants will be recruited through clinics. All the participants will be asked to keep a migraine diary for the duration of three months. In addition to that, the participants will fill out questionnaires that measures depression, anxiety, well-being and migraine related disability. This study does not intervene with the routine clinical care. The investigators merely observe through participant's diary and other patient reports to find out about how psychological and social factors might lead to different clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged between 18 and 65 who meet the International Headache Society's criteria for migraines

Exclusion Criteria:

* incapacitate such as dementia or cognitive deficiency
* illiterate, or could not sign informed consents
* severe disorder or co-morbidities that the doctors advice against participation

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: participants aged 18 to 65 who meet the International Headache Society's criteria for migraines.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-02-21 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Migraine attack frequency | 3 months
  The frequency of migraine attacks will be assessed by the number of days with migraine attacks recorded in the migraine diary.
Migraine attack intensity | 3 months
  The intensity of migraine attacks will be assessed by the Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst pain imaginable). Higher scores indicate greater pain intensity.
Migraine attack duration | 3 months
  The duration of each migraine attack will be recorded in the migraine diary, measured in hours.
Effectiveness of acute medication | 3 months
  The effectiveness of acute medication will be assessed by a 4-point scale measuring the degree of pain relief after medication administration, recorded in the migraine diary:
  1. No effect at all
  2. Minimal effect, headache slightly improved
  3. Good effect, headache significantly improved
  4. Very effective, pain completely resolved

SECONDARY OUTCOMES:
Compliance rate of migraine diary | 3 months
  The compliance rate of migraine diary will be calculated as the percentage of days with appropriately completed diary entries out of the total days of participation.
Compliance rate of lifestyle modification | 3 months
  The compliance rate of lifestyle modification will be assessed by self-reported adherence to recommended changes (e.g., sleeping time, or exercising) in the migraine diary.
depression | 3 months
  Depression will be assessed by the Patient Health Questionnaire-9 (PHQ-9). The scale ranges from 0 to 27, with higher scores indicating more severe depression.
anxiety | 3 months
  Anxiety will be assessed by the Generalized Anxiety Disorder-7 (GAD-7). The scale ranges from 0 to 21, with higher scores indicating more severe anxiety.
well-being | 3 months
  Well-being will be assessed by the Flourishing Scale. The scale ranges from 8 to 56, with higher scores indicating greater psychological well-being.
Pain Resilience | 3 months
  Pain resilience will be assessed by the Pain Resilience Scale (PRS). The scale ranges from 0 to 56, with higher scores indicating greater resilience to pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Chang-hua, Taiwan

IPD SHARING:
Plan to Share IPD: No
Since the research data contains medical records, we do not plan to share it.